CLINICAL TRIAL: NCT05790330
Title: 'Mind and Skin': A Prospective Cohort Study Evaluating the Impact of Inflammation, Itch and Sleep Disturbance on the Brain, Mental Health and Cognition, in Patients With Severe Atopy
Brief Title: Mind and Skin - the Neurocutaneous Axis in Atopic Eczema
Status: Recruiting | Type: Observational
Sponsor: King's College London (Other)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 280154
Record Dates: First submitted 2022-09-02; First posted 2023-03-30 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Methotrexate; dupilumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Severe eczema: Patients aged 12-18 who have been diagnosed with atopic eczema and require starting systemic therapy.
  Interventions: Drug: Methotrexate; Drug: Dupilumab
- Less severe eczema: Patients aged 12-18 who have been diagnosed with atopic eczema and require topical steroid therapy only.
- Healthy controls: Patients ages 12-18 who do not have atopic eczema.

INTERVENTIONS:
Drug: Methotrexate — As per usual standard of care
  Groups: Severe eczema
Drug: Dupilumab — As per usual standard of care
  Groups: Severe eczema

SUMMARY:
'Mind and Skin': A prospective cohort study evaluating the impact of inflammation, itch and sleep disturbance on the brain, mental health and cognition, in patients with severe atopy.

DETAILED DESCRIPTION:
Atopic eczema is an intensely itchy skin disease which often starts in infancy or early childhood. It can have profound effects on patients' quality of life and cause long-lasting psychological impairment. Sleep may be very disturbed. More severe disease often requires oral/injectable immuno-modulatory treatments (i.e. medications which control symptoms by influencing the immune system).

There is an association between eczema, impaired cognitive functioning and mental health disorders, but the underlying mechanisms are not clearly defined.

This projects examines the links between inflammation-driven itching and disturbed sleep, and how this might be causally responsible for systemic and brain inflammation, disturbance of cognitive functioning and mental health problems. The investigators will also study potential changes occurring following an improvement in eczema when patients are treated with systemic immuno-modulators.

Key investigations will include:

i) Home-based sleep studies using a commercially available sleep devices (for example DREEM headband, Philips Actiwatch, oximetry) ii) Structural and functional magnetic resonance imaging (MRI) of the brain, iii) Blood tests to quantify systemic inflammation iv) Genetic analyses, particularly related to the immune system, circadian rhythm (the "internal 24-hour clock"), skin barrier function and the risk of developing eczema or associated diseases, v) Assessments of the skin's barrier function vi) Stool samples and skin swabs to study the gut and skin microbiome.

The investigators will utilise existing anonymised data for comparative purposes (e.g. from patients with Attention Deficit Hyperactivity Disorder (ADHD) and healthy controls who previously had brain imaging.)

The investigators will explore eczema patients' and families' perception of their disease, in particular itch and the resulting sleep loss, through focus groups, to better understand the sociological impact of eczema, and how these patients' interactions with the external world and society are affected by eczema. Importantly, this will include exploration of family dynamics, as patients with eczema often have profound sleep disturbance from early life, which can impact on their caregivers' sleep and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 12 to 18 with atopic eczema (groups 1 and 2), which has been diagnosed by a Consultant Dermatologist.
2. Patients with atopic eczema warranting systemic immuno-modulatory therapy or patients with atopic eczema on topical therapy or healthy controls.
3. Written informed consent for study participation obtained from the patient or from the parent(s) / legal guardian, with assent as determined by the patient's age and level of understanding.
4. Willingness to comply with all study requirements.
5. Competent use of English language, according to patient's age (patients will be required to understand the written questionnaires and complying with instructions during MRI scanning).

Exclusion Criteria:

1. Insufficient understanding of the study by the patient and/or parent/guardian.
2. Any clear contra-indication to MRI scanning. In particular this would be due to the presence of any implanted devices or metal from previous surgery or accident. This would be fully assessed with a standardised safety questionnaire by a radiographer prior to MRI scanning.
3. Any condition deemed by the Investigator to limit a patient's ability to undertake MRI components of the study, for example significant claustrophobia.
4. Diagnosed by a sleep medicine specialist with a formal sleep disorder, requiring systemic medication.
5. Sleep disturbance from co-morbid illness (including physical and/or mental/psychological illness) other than atopic eczema, deemed by the Investigator to significantly impact on sleep components of the study.
6. Previous and/or current substance misuse.
7. Patients who take medications that would, in the investigator's opinion, impact on quality of sleep studies.

Ages: 12 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Group 1: Patients aged 12-18 who have been diagnosed with eczema and require systemic therapy.
  Group 2: Patients aged 12-18 who have been diagnosed with eczema and require topical therapy only.
  Group 3: Patients aged 12-18 who do not have eczema.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2023-03-10 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Eczema Area and Severity Index (EASI) Score | 6 months
  Clinical assessment of atopic dermatitis disease activity. Range 0-72 (72 being the most severe outcome)
Peak Pruritus Numerical Rating Score | 6 months
  Patient reported itch severity. Range 0-10 (10 being the worst outcome)
Transepidermal water loss (TEWL) | 6 months
  Skin barrier function measurement using a device which measures the amount of water that passively evaporates through skin to the external environment due to water vapor pressure gradient on both sides of the skin barrier
Skin surface pH | 6 months
  Skin barrier function measurement using a pH measuring device.
Metabolome swab | 6 months
  Skin metabalome analysis using a skin swab
Skin ELISA (enzyme-linked immunosorbent assay) and serum ELISA | 6 months
  Immunoassay detection and quantification
RNA sequencing of blood serum | 6 months
  To detect transcript isoforms, gene fusions and single nucleotide variants.
Pediatric Sleep Questionnaire | 6 months
  Sleep questionnaire. Score 18-126 (126 being the worst clinical outcome)
Morningness-Eveningness Questionnaire | 6 months
  Sleep questionnaire. Score 16-86 assesses individual differences in morningness and eveningness - the degree to which respondents are active and alert at certain times of day.
Patient-Reported Outcomes Measurement Information System (PROMIS) | 6 months
  Sleep questionnaire. Score 0-20 (0 being the worst clinical outcome)
Pittsburgh Sleep Quality Index | 6 months
  Sleep questionnaires. Score 0-21 (21 being the worst clinical outcome)
Dreem headband electroencephalogram monitoring | 6 months
  Sleep study - Measures brain activity to assess sleep cycles
Polysomnography | 6 months
  Sleep study incorporating electroencephalogram, electro-oculogram, electromyogram, electrocardiogram, and pulse oximetry, as well as airflow and respiratory effort, to evaluate for underlying causes of sleep disturbances.
Actigraphy Watch analysis | 6 months
  Watch is worn by participant which records movement during sleep to analyse sleep pattern
EMFIT mattress analysis | 6 months
  Mattress sensor which records movement during sleep to analyse sleep pattern to analyse sleep pattern
Wechsler Abbreviated Scale of Intelligence Second Edition (WASI-II) Score | 6 months
  Intelligence Quotient Test. Score 40-160 (40 being the worst clinical outcome)
Go/No-GO Task | 6 months
  The Go/No-go task requires participants to respond by pressing a button when they see a "go" signal, and not respond when they see the "no-go" signal. The key behaviour measured with this experiment is the participants' ability to withhold a response on No-go trials. This is scored as a fraction of correct responses.
Simon Task | 6 months
  In this task participants are asked to respond to visual stimuli by making a rightward response to one stimulus (e.g. a circle) and a leftward response to another (e.g. a square). This is scored as a fraction of correct responses.
Continuous Performance Task | 6 months
  In this task participants are asked to only respond to a specific sequence of visual stimuli. This is scored as a fraction of correct responses.
Time Discrimination Task | 6 months
  In this task participants are ask to decide which stimuli stayed on screen for the longest duration. This is scored as a fraction of correct responses.
Vigilance Task (Mackworth Clock) | 6 months
  In this task participants are asked to watched a clock hand that moves every second around the clock. From time to time the hand skips a second and participants need to respond to this. This is scored as a fraction of correct responses.
Performance on Working Memory Task | 6 months
  Completed in functional MRI
Performance on Sustained Attention Task | 6 months
  Completed in functional MRI
Resting Brain State | 6 months
  Measured in functional MRI
Structural Changes in the Brain | 6 months
  Structure of the brain is measured in MRI

CONTACTS AND LOCATIONS:
Locations (1):
- Unit for Paediatric and Population-based Dermatology Research, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No